CLINICAL TRIAL: NCT02431520
Title: Patient Compliance to Self-collection for Detection of HPV-DNA in Cervical Cancer Prevention: A Clinical Trial
Brief Title: Patient Compliance to Self-collection for Detection of HPV-DNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 58/07
Record Dates: First submitted 2014-09-15; First posted 2015-05-01 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Compliance; Cervical Cancer
Keywords: Patient Compliance; HPV-DNA probes; Papanicolaou test; Cervical cancer
MeSH Terms: conditions — Patient Compliance; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-collection (Experimental): Women allocated to this arm will be asked to obtain a specimen of vaginal/cervical by self-collection for Hybrid Capture II (HCII).
  Interventions: Procedure: Self-collection
- Gynecologist collection (Active Comparator): Women allocated to this arm will be asked to attend to medical office to have their Pap smear obtained by a gynecologist
  Interventions: Procedure: Gynecologist collection

INTERVENTIONS:
Procedure: Self-collection — Women allocated to this arm will be asked to obtain a specimen of vaginal/cervical by self-collection for HCII.
  Arms: Self-collection
Procedure: Gynecologist collection — Women allocated to this arm will be asked to attend to medical office to have their Pap smear obtained by a gynecologist
  Arms: Gynecologist collection

SUMMARY:
A study to investigate the compliance of unassisted women to self-collection of specimens for Hybrid Capture (HC) for detection of Human Papilloma Virus (HPV) DNA compared to Pap smear collection by medical personnel, as screening method to identify precursor lesions of cervical cancer.

DETAILED DESCRIPTION:
Women living in the community of the Morro dos Macacos, Vila Isabel, Rio de Janeiro, were randomly allocated for self-collection of specimens for HC II for detection of HPV-DNA or to Pap smear collection by medical personnel, as screening method to identify precursor lesions of cervical cancer.

The compliance was measured by the delivery of the specimen obtained by self-collection or to attend to a visit at the community health center to be submitted to Pap smear collection, within a week.

ELIGIBILITY:
Inclusion Criteria:

* Women between 25-59 years-old
* Not pregnant
* Had held their last Pap smear for over a year
* Could read.

Exclusion Criteria:

* Women with previous hysterectomy
* History of cervical cancer or its precursors
* Bearers of some state of chronic immunosuppression (such as HIV ou autoimmune diseases)
* Those who underwent self-collection of their specimen during menstrual period

Ages: 25 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Compliance to self-collection for detection of HPV-DNA measured by the percentage of subjects that returned the vaginal self-collected sample or attended to the medical appointment according to allocation. | One week after inclusion
  Risk of compliance to self-collection for detection of HPV-DNA in relation to collection by medical personnel

CONTACTS AND LOCATIONS:
Overall Officials: Fabio B Russomano, MD, PhD, Principal Investigator — IFF/Fiocruz
Locations (1):
- Instituto Nacional de Saúde da Mulher, da Criança e do Adolescente Fernandes Figueira (IFF/Fiocruz), Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Brink AA, Meijer CJ, Wiegerinck MA, Nieboer TE, Kruitwagen RF, van Kemenade F, Fransen Daalmeijer N, Hesselink AT, Berkhof J, Snijders PJ. High concordance of results of testing for human papillomavirus in cervicovaginal samples collected by two methods, with comparison of a novel self-sampling device to a conventional endocervical brush. J Clin Microbiol. 2006 Jul;44(7):2518-23. doi: 10.1128/JCM.02440-05. PMID 16825374
- [Background] Cuzick J. Human papillomavirus testing for primary cervical cancer screening. JAMA. 2000 Jan 5;283(1):108-9. doi: 10.1001/jama.283.1.108. No abstract available. PMID 10632290
- [Background] Dzuba IG, Diaz EY, Allen B, Leonard YF, Lazcano Ponce EC, Shah KV, Bishai D, Lorincz A, Ferris D, Turnbull B, Hernandez Avila M, Salmeron J. The acceptability of self-collected samples for HPV testing vs. the pap test as alternatives in cervical cancer screening. J Womens Health Gend Based Med. 2002 Apr;11(3):265-75. doi: 10.1089/152460902753668466. PMID 11988136
- [Background] Gontijo RC, Derchain SF, Montemor EB, Sarian LO, Serra MM, Zeferino LC, Syrjanen KJ. [Pap smear, hybrid capture II, and visual inspection in screening for uterine cervical lesions]. Cad Saude Publica. 2005 Jan-Feb;21(1):141-9. doi: 10.1590/s0102-311x2005000100016. Epub 2005 Jan 28. Portuguese. PMID 15692647
- [Background] Harper DM, Hildesheim A, Cobb JL, Greenberg M, Vaught J, Lorincz AT. Collection devices for human papillomavirus. J Fam Pract. 1999 Jul;48(7):531-5. PMID 10428251
- [Background] Wikstrom I, Stenvall H, Wilander E. Attitudes to self-sampling of vaginal smear for human papilloma virus analysis among women not attending organized cytological screening. Acta Obstet Gynecol Scand. 2007;86(6):720-5. doi: 10.1080/00016340701303747. PMID 17520406
- [Background] Wright TC Jr, Denny L, Kuhn L, Pollack A, Lorincz A. HPV DNA testing of self-collected vaginal samples compared with cytologic screening to detect cervical cancer. JAMA. 2000 Jan 5;283(1):81-6. doi: 10.1001/jama.283.1.81. PMID 10632284
- [Background] Mandelblatt JS, Lawrence WF, Womack SM, Jacobson D, Yi B, Hwang YT, Gold K, Barter J, Shah K. Benefits and costs of using HPV testing to screen for cervical cancer. JAMA. 2002 May 8;287(18):2372-81. doi: 10.1001/jama.287.18.2372. PMID 11988058
- [Background] Ogilvie G, Krajden M, Maginley J, Isaac-Renton J, Hislop G, Elwood-Martin R, Sherlock C, Taylor D, Rekart M. Feasibility of self-collection of specimens for human papillomavirus testing in hard-to-reach women. CMAJ. 2007 Aug 28;177(5):480-3. doi: 10.1503/cmaj.070013. PMID 17724326